CLINICAL TRIAL: NCT05704725
Title: An Open Label, Two-Arm Study in Subjects With Chorioretinal Vascular Disease to Evaluate ABP 938 and Aflibercept (Eylea®) in a Prefilled Syringe
Brief Title: A Study to Evaluate ABP 938 and Aflibercept (Eylea®) in Participants With Chorioretinal Vascular Disease (CVD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210034; 2019-002503-17 (EudraCT Number)
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Chorioretinal Vascular Disease
Keywords: Chorioretinal vascular disease; CVD; ABP 938; EYLEA®; aflibercept
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ABP 938 (Experimental): Participants will be randomized in a ratio of 2:1 to receive either a single IVT injection of ABP 938 in a PFS or a single injection of aflibercept in a PFS.
  Interventions: Drug: ABP 938
- Aflibercept (Experimental): Participants will be randomized in a ratio of 2:1 to receive either a single IVT injection of ABP 938 in a PFS or a single injection of aflibercept in a PFS.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: ABP 938 — IVT injection
  Other Names: PAVBLU™
  Arms: ABP 938
Drug: Aflibercept — IVT injection
  Other Names: Eylea®
  Arms: Aflibercept

SUMMARY:
The primary objective of this study is to is to assess the ability of retina specialists to successfully administer, via an intravitreal (IVT) injection, a 2 mg dose of ABP 938, using the ABP 938 aflibercept prefilled syringe (PFS), compared to a 2 mg dose of aflibercept using the aflibercept PFS.

ELIGIBILITY:
Inclusion Criteria

* Must sign an IRB approved informed consent form before any study-specific procedures are initiated.
* Men or women ≥18 years old.
* Treatment-naïve or previously treated neovascular age-related macular degeneration, diabetic macular edema, macular edema following retinal vein occlusion, or diabetic retinopathy in the study eye.

Exclusion Criteria

* Active intraocular or periocular infection or active intraocular inflammation in either eye.
* Uncontrolled intraocular pressure greater than (>) 25 mmHg in the study eye.
* Deemed legally blind in one or both eyes.
* History of or any current indication of excessive bleeding or recurrent hemorrhages, including any prior excessive intraocular bleeding or hemorrhages after IVT injection or intraocular procedures in either eye.
* Current systemic infectious disease or on a therapy for active infectious disease.
* History of any medical, ocular or non-ocular conditions that, in the opinion of the investigator, may interfere with the injection procedure or pose a safety concern.
* History of stroke or transient ischemic attacks or myocardial infarction within the last 6 months.
* Treatment with anti-VEGF IVT injection in the study eye within 28 days.
* Any use of intraocular corticosteroids in the study eye within 3 months.
* Receipt of any systemic anti-VEGF within the last 6 months.
* Any invasive intraocular surgery, prior long-acting therapeutic agent, or ocular drug release device implantation in the study eye within the past 3 months.
* For women: pregnant or breast feeding, or planning to become pregnant while enrolled in the study and for 3 months after IP administration.
* Sexually active participants and their partners who are of childbearing potential who refuse to use adequate contraception while on-study and for 3 months after IP administration. Male participants must agree not to donate sperm during study and for 3 months following dose of IP.
* Allergy or hypersensitivity to the IP, to any of the excipients of ABP 938 or aflibercept, or to other study-related procedures/medications.
* Previously enrolled in this study.
* Participation in any interventional clinical study within 3 months prior to screening.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- United States (4):
  - Retina Consultants of Texas - Austin Retina, Austin, Texas
  - Retina Consultants of Texas - Bellaire Retina Center, Bellaire, Texas
  - Retinal Consultants of Texas - San Antonio Retina Center, San Antonio, Texas
  - Retina Consultants of Texas - The Woodlands Retina Center, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 4 centers in the United States between 23 January 2023 and 24 March 2023.
Pre-assignment Details: Participants were randomized in a ratio of 2:1 to receive either a single intravitreal (IVT) injection of ABP 938 in a pre-filled syringe (PFS) or a single injection of aflibercept in a PFS.
Groups:
- ABP 938: Participants received a single 2.0 mg/0.05 mL IVT injection of ABP 938 by PFS.
- Aflibercept: Participants received a single 2.0 mg/0.05 mL IVT injection of aflibercept by PFS.
Period: Overall Study
Arm/Group | ABP 938 | Aflibercept
Started | 33 | 16
Completed | 32 | 15
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | ABP 938 | Aflibercept | Total
Number analyzed (Participants) | 33 | 16 | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.0 (11.40) | 66.3 (15.64) | 69.5 (12.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 2 | 16
  Male | 19 | 14 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 4 | 13
  Not Hispanic or Latino | 23 | 12 | 35
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 28 | 14 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of IVT Injections Successfully Administered
Description: A successful injection was defined by whether the retinal specialist administering the IVT injection answered 'yes' to the following question: Did the PFS allow for the safe and effective administration of the prescribed dose? Percentage of successful injections and Clopper-Pearson 95% Confidence Interval is reported.
Time Frame: Day of IVT injection (study day 1)
Population: FAS (only participants with available data are included.)
Measure: Number (95% Confidence Interval); unit: Percentage of Successful Injections
Arm/Group | ABP 938 | Aflibercept
Number analyzed (Participants) | 32 | 16
Percentage of Successful Injections | 100 [89.1 to 100.0] | 100 [79.4 to 100.0]

2. Secondary Outcome: Number of Participants With Ocular Treatment Emergent Adverse Events (TEAEs) in Study Eye
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant. Events that met the AE definition are as follows:
  * Any abnormal or worsening ocular safety result that is considered clinically significant in the medical and scientific judgment of the investigator.
  * Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition.
  * New conditions detected or diagnosed after study treatment administration even though it may have been present before the start of the study.
  * Signs, symptoms, or the clinical sequelae of a suspected overdose of either study treatment or a concomitant medication.
  AEs were classified by system organ class (SOC) according to the Medical Dictionary for Regulatory Activities (medDRA) and graded by Common Terminology Criteria for Adverse Events (CTCAE), version 5.0
Time Frame: Up to 28 days
Population: Safety Analysis Set (SAS): all randomized participants who received investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | ABP 938 | Aflibercept
Number analyzed (Participants) | 32 | 16
Participants | 3 | 0

3. Secondary Outcome: Number of Participants With Serious Ocular TEAEs in Study Eye
Description: A serious AE is any event that met at least 1 of the following serious criteria:
  * Fatal.
  * Life-threatening (places the participant at immediate risk of death).
  * Requires inpatient hospitalization or prolongation of existing hospitalization.
  * Results in persistent or significant disability/incapacity.
  * Congenital anomaly/birth defect.
  * Other medically important serious event.
  AEs were classified by SOC according to medDRA and graded by CTCAE, version 5.0
Time Frame: Up to 28 days
Population: SAS
Measure: Count of Participants; unit: Participants
Arm/Group | ABP 938 | Aflibercept
Number analyzed (Participants) | 32 | 16
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Non-ocular Serious TEAEs
Description: as for outcome 3
Time Frame: Up to 28 days
Population: SAS
Measure: Count of Participants; unit: Participants
Arm/Group | ABP 938 | Aflibercept
Number analyzed (Participants) | 32 | 16
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | ABP 938 | Aflibercept
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/16
Other Adverse Events (participants affected / at risk) | 2/32 | 2/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABP 938 (N=32) | Aflibercept (N=16)
Vitreous detachment (Eye disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT05704725/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT05704725/SAP_001.pdf